CLINICAL TRIAL: NCT05392959
Title: Effect of the Antidiabetic Drug DAPAgliflozin on the Coronary Macrovascular and MICROvascular Function in Type 2 Diabetic Patients
Acronym: DAPAMICRO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment too slow
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B0762021210908
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Dapagliflozin; Physiological Effects of Drugs; Coronary Artery Disease; Microcirculation; Fraction Flow Reserve; Index of Microcirculatory Resistance; Coronary Flow Reserve
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): The patient will be treated in standard of care for type 2 diabetic mellitus and will receive a placebo (1 tablet) administered orally daily during 24 weeks
  Interventions: Drug: Placebo
- dapagliflozin group (Experimental): The patient will be treated in standard of care for type 2 diabetic mellitus and will receive Dapagliflozin 10 mg (1 tablet) administered orally daily during 24 weeks
  Interventions: Drug: Dapagliflozin 10 mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10 mg Tab — Dapagliflozin 10 mg per day
  Other Names: Forxiga®
  Arms: dapagliflozin group
Drug: Placebo — Placebo for dapagliflozin film-coated tablets 10 mg
  Arms: Placebo group

SUMMARY:
Cardiovascular events remain a major driver of morbidity and mortality in patients with type 2 diabetes mellitus. Diffuse coronary atherosclerosis, combined with impairment of the microcirculation are frequent even in asymptomatic patients and can lead to unfavourable outcomes. In recent years, novel classes of antidiabetic drugs have been introduced, with salutary effects on cardiovascular outcomes of diabetic patients. The sodium-glucose linked transporter 2 (SGLT2) inhibitors - gliflozins - bind to the SGLT2 receptors of the proximal tubule of the nephron and cause glycosuria. They have been shown to have favourable cardiovascular effects by reducing deaths from cardiovascular causes in type 2 diabetic patients.

Moreover, dapagliflozin reduces hospitalisation for heart failure in type 2 diabetic heart failure patients with and without reduced ejection fraction and reduces cardiovascular death and all causes mortality in those with reduced ejection fraction.

It is currently unknown if this is mediated by improvement of coronary physiology both at the level of the epicardial coronary arteries as well as the coronary microcirculation.

The purpose of the study is to explore the impact of dapagliflozin on the coronary and microcirculatory function of type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus (T2DM) patients presenting with stable angina and a clinical indication for cardiac catheterization
* T2DM patients with non ST elevation myocardial infarction (NSTEMI) or unstable angina referred for cardiac catheterization
* Demonstration of coronary lesion(s) with non-significant fractional flow reserve (FFR) values (>0.80), for which revascularisation is deferred
* Agreement to practice an acceptable method of birth control for women of childbearing potential
* Signed patient informed consent

Exclusion Criteria:

* Age < 18 years old
* T2DM patients presenting with ST elevation myocardial infarction (STEMI)
* Pregnancy or breastfeeding
* Body mass index ≥45 kg/m2
* Creatinine clearance ≤45 ml/min/1.73 m2 (as calculated by Modification of Diet in Renal Disease Study (MDRD ) formula for estimated Glomerular filtration rate (GFR))
* Indication of liver disease, defined by serum levels of alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase above 3 x upper limit of normal during screening or run-in phase
* Uncontrolled hyperglycemia with glucose >240 mg/dL after an overnight fast
* Stroke, or transient ischemic attack at presentation and up to 2 months prior to informed consent
* Alcohol or drug abuse within 3 months of informed consent that would interfere with trial participation or any ongoing condition leading to decreased compliance with study procedures or study drug intake
* Any uncontrolled endocrine disorder except type 2 diabetes
* Treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent
* Treatment with anti-obesity drugs 3 months prior to informed consent or any other treatment at time of screening leading to unstable body weight
* Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years
* Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells
* Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption
* Planned cardiac surgery or angioplasty within 3 months
* Any clinical condition that would jeopardize patient safety while participating in this clinical trial
* Life expectancy < 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
the longitudinal change of the Fractional Flow Reserve (FRR) | up to 6 months
  The longitudinal change (Δ) of FFR is defined as the value at follow-up (6 months) minus the value at baseline.
  The complete assessment of the function of the coronary circulation will be performed by using a dedicated pressure and temperature equipped coronary guidewire (PressureWire X by Abbott Vascular) and the Coroventis CoroFlow software platform.
  In the presence of coronary lesions, the degree of percent diameter stenosis will be measured by quantitative coronary angiography and their hemodynamic significance will be evaluated by measuring fractional flow reserve (FFR). According to the guidelines for myocardial revascularisation, only the lesions that have an FFR value equal or less than 0.8 will be treated by coronary angioplasty . In case of angioplasty, FFR will be also measured immediately after successful implantation of the coronary stent.
the longitudinal change of the Coronary flow reserve (CFR) | up to 6 months
  The longitudinal change (Δ) of CFR is defined as the value at follow-up (6 months) minus the value at baseline.
  The complete assessment of the function of the coronary circulation will be performed by using a dedicated pressure and temperature equipped coronary guidewire (PressureWire X by Abbott Vascular) and the Coroventis CoroFlow software platform.
  Coronary flow reserve (CFR) will be measured in the vessels of interest, where FFR was measured.
the longitudinal change of the Index of Microvascular Resistance (IMR). | up to 6 months
  The longitudinal change (Δ) of IMR is defined as the value at follow-up (6 months) minus the value at baseline.
  The complete assessment of the function of the coronary circulation will be performed by using a dedicated pressure and temperature equipped coronary guidewire (PressureWire X by Abbott Vascular) and the Coroventis CoroFlow software platform.
  The Index of Microvascular Resistance (IMR) will be measured in the vessels of interest, where FFR was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Xaplanteris, MD, PhD, Principal Investigator — panagiotis.xaplanteris@stpierre-bru.be
Locations (1):
- CHU Saint Pierre, Brussels, Bruxelles-Capitale, Région de;Brussels Hoofdstedelijk Gewest, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrannini E, Ramos SJ, Salsali A, Tang W, List JF. Dapagliflozin monotherapy in type 2 diabetic patients with inadequate glycemic control by diet and exercise: a randomized, double-blind, placebo-controlled, phase 3 trial. Diabetes Care. 2010 Oct;33(10):2217-24. doi: 10.2337/dc10-0612. Epub 2010 Jun 21. PMID 20566676
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR. Management of hyperglycemia in type 2 diabetes, 2015: a patient-centered approach: update to a position statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2015 Jan;38(1):140-9. doi: 10.2337/dc14-2441. No abstract available. PMID 25538310
- [Background] DeFronzo RA, Norton L, Abdul-Ghani M. Renal, metabolic and cardiovascular considerations of SGLT2 inhibition. Nat Rev Nephrol. 2017 Jan;13(1):11-26. doi: 10.1038/nrneph.2016.170. Epub 2016 Dec 12. PMID 27941935
- [Background] Bailey CJ, Gross JL, Pieters A, Bastien A, List JF. Effect of dapagliflozin in patients with type 2 diabetes who have inadequate glycaemic control with metformin: a randomised, double-blind, placebo-controlled trial. Lancet. 2010 Jun 26;375(9733):2223-33. doi: 10.1016/S0140-6736(10)60407-2. PMID 20609968
- [Background] Wilding JP, Rajeev SP, DeFronzo RA. Positioning SGLT2 Inhibitors/Incretin-Based Therapies in the Treatment Algorithm. Diabetes Care. 2016 Aug;39 Suppl 2:S154-64. doi: 10.2337/dcS15-3005. PMID 27440828
- [Background] Abdul-Ghani M, Del Prato S, Chilton R, DeFronzo RA. SGLT2 Inhibitors and Cardiovascular Risk: Lessons Learned From the EMPA-REG OUTCOME Study. Diabetes Care. 2016 May;39(5):717-25. doi: 10.2337/dc16-0041. PMID 27208375
- [Background] Zhou H, Wang S, Zhu P, Hu S, Chen Y, Ren J. Empagliflozin rescues diabetic myocardial microvascular injury via AMPK-mediated inhibition of mitochondrial fission. Redox Biol. 2018 May;15:335-346. doi: 10.1016/j.redox.2017.12.019. Epub 2017 Dec 30. PMID 29306791
- [Background] Ott C, Jumar A, Striepe K, Friedrich S, Karg MV, Bramlage P, Schmieder RE. A randomised study of the impact of the SGLT2 inhibitor dapagliflozin on microvascular and macrovascular circulation. Cardiovasc Diabetol. 2017 Feb 23;16(1):26. doi: 10.1186/s12933-017-0510-1. PMID 28231831
- [Background] van Bommel EJM, Muskiet MHA, Tonneijck L, Kramer MHH, Nieuwdorp M, van Raalte DH. SGLT2 Inhibition in the Diabetic Kidney-From Mechanisms to Clinical Outcome. Clin J Am Soc Nephrol. 2017 Apr 3;12(4):700-710. doi: 10.2215/CJN.06080616. Epub 2017 Mar 2. PMID 28254770
- [Background] Scheen AJ. Pharmacodynamics, efficacy and safety of sodium-glucose co-transporter type 2 (SGLT2) inhibitors for the treatment of type 2 diabetes mellitus. Drugs. 2015 Jan;75(1):33-59. doi: 10.1007/s40265-014-0337-y. PMID 25488697
- [Background] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Background] Kato ET, Silverman MG, Mosenzon O, Zelniker TA, Cahn A, Furtado RHM, Kuder J, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Bonaca MP, Ruff CT, Desai AS, Goto S, Johansson PA, Gause-Nilsson I, Johanson P, Langkilde AM, Raz I, Sabatine MS, Wiviott SD. Effect of Dapagliflozin on Heart Failure and Mortality in Type 2 Diabetes Mellitus. Circulation. 2019 May 28;139(22):2528-2536. doi: 10.1161/CIRCULATIONAHA.119.040130. Epub 2019 Mar 18. PMID 30882238
- [Background] Kolh P, Windecker S, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A; European Society of Cardiology Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; EACTS Clinical Guidelines Committee; Sousa Uva M, Achenbach S, Pepper J, Anyanwu A, Badimon L, Bauersachs J, Baumbach A, Beygui F, Bonaros N, De Carlo M, Deaton C, Dobrev D, Dunning J, Eeckhout E, Gielen S, Hasdai D, Kirchhof P, Luckraz H, Mahrholdt H, Montalescot G, Paparella D, Rastan AJ, Sanmartin M, Sergeant P, Silber S, Tamargo J, ten Berg J, Thiele H, van Geuns RJ, Wagner HO, Wassmann S, Wendler O, Zamorano JL; Task Force on Myocardial Revascularization of the European Society of Cardiology and the European Association for Cardio-Thoracic Surgery; European Association of Percutaneous Cardiovascular Interventions. 2014 ESC/EACTS Guidelines on myocardial revascularization: the Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur J Cardiothorac Surg. 2014 Oct;46(4):517-92. doi: 10.1093/ejcts/ezu366. Epub 2014 Aug 29. No abstract available. PMID 25173601
- [Background] Gould KL, Lipscomb K, Hamilton GW. Physiologic basis for assessing critical coronary stenosis. Instantaneous flow response and regional distribution during coronary hyperemia as measures of coronary flow reserve. Am J Cardiol. 1974 Jan;33(1):87-94. doi: 10.1016/0002-9149(74)90743-7. No abstract available. PMID 4808557
- [Background] Barbato E, Aarnoudse W, Aengevaeren WR, Werner G, Klauss V, Bojara W, Herzfeld I, Oldroyd KG, Pijls NH, De Bruyne B; Week 25 study group. Validation of coronary flow reserve measurements by thermodilution in clinical practice. Eur Heart J. 2004 Feb;25(3):219-23. doi: 10.1016/j.ehj.2003.11.009. PMID 14972422
- [Background] Cortigiani L, Rigo F, Gherardi S, Galderisi M, Bovenzi F, Picano E, Sicari R. Prognostic effect of coronary flow reserve in women versus men with chest pain syndrome and normal dipyridamole stress echocardiography. Am J Cardiol. 2010 Dec 15;106(12):1703-8. doi: 10.1016/j.amjcard.2010.08.011. PMID 21126613
- [Background] Johnson NP, Kirkeeide RL, Gould KL. Is discordance of coronary flow reserve and fractional flow reserve due to methodology or clinically relevant coronary pathophysiology? JACC Cardiovasc Imaging. 2012 Feb;5(2):193-202. doi: 10.1016/j.jcmg.2011.09.020. PMID 22340827
- [Background] Meuwissen M, Chamuleau SA, Siebes M, Schotborgh CE, Koch KT, de Winter RJ, Bax M, de Jong A, Spaan JA, Piek JJ. Role of variability in microvascular resistance on fractional flow reserve and coronary blood flow velocity reserve in intermediate coronary lesions. Circulation. 2001 Jan 16;103(2):184-7. doi: 10.1161/01.cir.103.2.184. PMID 11208673
- [Background] Pijls NH, van Son JA, Kirkeeide RL, De Bruyne B, Gould KL. Experimental basis of determining maximum coronary, myocardial, and collateral blood flow by pressure measurements for assessing functional stenosis severity before and after percutaneous transluminal coronary angioplasty. Circulation. 1993 Apr;87(4):1354-67. doi: 10.1161/01.cir.87.4.1354. PMID 8462157
- [Background] De Bruyne B, Baudhuin T, Melin JA, Pijls NH, Sys SU, Bol A, Paulus WJ, Heyndrickx GR, Wijns W. Coronary flow reserve calculated from pressure measurements in humans. Validation with positron emission tomography. Circulation. 1994 Mar;89(3):1013-22. doi: 10.1161/01.cir.89.3.1013. PMID 8124786
- [Background] Topol EJ, Ellis SG, Cosgrove DM, Bates ER, Muller DW, Schork NJ, Schork MA, Loop FD. Analysis of coronary angioplasty practice in the United States with an insurance-claims data base. Circulation. 1993 May;87(5):1489-97. doi: 10.1161/01.cir.87.5.1489. PMID 8141866
- [Background] De Bruyne B, Hersbach F, Pijls NH, Bartunek J, Bech JW, Heyndrickx GR, Gould KL, Wijns W. Abnormal epicardial coronary resistance in patients with diffuse atherosclerosis but "Normal" coronary angiography. Circulation. 2001 Nov 13;104(20):2401-6. doi: 10.1161/hc4501.099316. PMID 11705815
- [Background] De Bruyne B, Pijls NH, Paulus WJ, Vantrimpont PJ, Sys SU, Heyndrickx GR. Transstenotic coronary pressure gradient measurement in humans: in vitro and in vivo evaluation of a new pressure monitoring angioplasty guide wire. J Am Coll Cardiol. 1993 Jul;22(1):119-26. doi: 10.1016/0735-1097(93)90825-l. PMID 8509531
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] De Bruyne B, Fearon WF, Pijls NH, Barbato E, Tonino P, Piroth Z, Jagic N, Mobius-Winckler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd K, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Limacher A, Nuesch E, Juni P; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI for stable coronary artery disease. N Engl J Med. 2014 Sep 25;371(13):1208-17. doi: 10.1056/NEJMoa1408758. Epub 2014 Sep 1. PMID 25176289
- [Background] Pijls NH, De Bruyne B, Peels K, Van Der Voort PH, Bonnier HJ, Bartunek J Koolen JJ, Koolen JJ. Measurement of fractional flow reserve to assess the functional severity of coronary-artery stenoses. N Engl J Med. 1996 Jun 27;334(26):1703-8. doi: 10.1056/NEJM199606273342604. PMID 8637515
- [Background] Pijls NH, Van Gelder B, Van der Voort P, Peels K, Bracke FA, Bonnier HJ, el Gamal MI. Fractional flow reserve. A useful index to evaluate the influence of an epicardial coronary stenosis on myocardial blood flow. Circulation. 1995 Dec 1;92(11):3183-93. doi: 10.1161/01.cir.92.11.3183. PMID 7586302
- [Background] De Bruyne B, Pijls NH, Bartunek J, Kulecki K, Bech JW, De Winter H, Van Crombrugge P, Heyndrickx GR, Wijns W. Fractional flow reserve in patients with prior myocardial infarction. Circulation. 2001 Jul 10;104(2):157-62. doi: 10.1161/01.cir.104.2.157. PMID 11447079
- [Background] Xaplanteris P, Fournier S, Pijls NHJ, Fearon WF, Barbato E, Tonino PAL, Engstrom T, Kaab S, Dambrink JH, Rioufol G, Toth GG, Piroth Z, Witt N, Frobert O, Kala P, Linke A, Jagic N, Mates M, Mavromatis K, Samady H, Irimpen A, Oldroyd K, Campo G, Rothenbuhler M, Juni P, De Bruyne B; FAME 2 Investigators. Five-Year Outcomes with PCI Guided by Fractional Flow Reserve. N Engl J Med. 2018 Jul 19;379(3):250-259. doi: 10.1056/NEJMoa1803538. Epub 2018 May 22. PMID 29785878
- [Background] Fearon WF, Balsam LB, Farouque HM, Caffarelli AD, Robbins RC, Fitzgerald PJ, Yock PG, Yeung AC. Novel index for invasively assessing the coronary microcirculation. Circulation. 2003 Jul 1;107(25):3129-32. doi: 10.1161/01.CIR.0000080700.98607.D1. Epub 2003 Jun 23. PMID 12821539
- [Background] De Bruyne B, Barbato E. Quantitative assessment of the coronary microvasculature: new tools for the black box. Circulation. 2013 Jun 18;127(24):2378-9. doi: 10.1161/CIRCULATIONAHA.113.003361. Epub 2013 May 16. No abstract available. PMID 23681065
- [Background] Fearon WF, Low AF, Yong AS, McGeoch R, Berry C, Shah MG, Ho MY, Kim HS, Loh JP, Oldroyd KG. Prognostic value of the Index of Microcirculatory Resistance measured after primary percutaneous coronary intervention. Circulation. 2013 Jun 18;127(24):2436-41. doi: 10.1161/CIRCULATIONAHA.112.000298. Epub 2013 May 16. PMID 23681066
- [Background] Aarnoudse W, Fearon WF, Manoharan G, Geven M, van de Vosse F, Rutten M, De Bruyne B, Pijls NH. Epicardial stenosis severity does not affect minimal microcirculatory resistance. Circulation. 2004 Oct 12;110(15):2137-42. doi: 10.1161/01.CIR.0000143893.18451.0E. Epub 2004 Oct 4. PMID 15466646
- [Background] Ng MK, Yong AS, Ho M, Shah MG, Chawantanpipat C, O'Connell R, Keech A, Kritharides L, Fearon WF. The index of microcirculatory resistance predicts myocardial infarction related to percutaneous coronary intervention. Circ Cardiovasc Interv. 2012 Aug 1;5(4):515-22. doi: 10.1161/CIRCINTERVENTIONS.112.969048. Epub 2012 Aug 8. PMID 22874078
- [Background] Hennigan B, Layland J, Fearon WF, Oldroyd KG. Fractional flow reserve and the index of microvascular resistance in patients with acute coronary syndromes. EuroIntervention. 2014 Aug;10 Suppl T:T55-63. doi: 10.4244/EIJV10STA10. PMID 25256535
- [Background] Xaplanteris P, Ntalianis A, De Bruyne B, Strisciuglio T, Pellicano M, Ciccarelli G, Milkas A, Barbato E. Coronary lesion progression as assessed by fractional flow reserve (FFR) and angiography. EuroIntervention. 2018 Oct 20;14(8):907-914. doi: 10.4244/EIJ-D-17-00872. PMID 29769166
- [Background] Zimmermann FM, Ferrara A, Johnson NP, van Nunen LX, Escaned J, Albertsson P, Erbel R, Legrand V, Gwon HC, Remkes WS, Stella PR, van Schaardenburgh P, Bech GJ, De Bruyne B, Pijls NH. Deferral vs. performance of percutaneous coronary intervention of functionally non-significant coronary stenosis: 15-year follow-up of the DEFER trial. Eur Heart J. 2015 Dec 1;36(45):3182-8. doi: 10.1093/eurheartj/ehv452. Epub 2015 Sep 23. PMID 26400825